CLINICAL TRIAL: NCT03104582
Title: Best Biliary Drainage Option in Type II、III、IV Klatskin Tumor：ERCP or PTBD
Brief Title: Best Biliary Drainage Option in Advanced Klatskin Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, M.D., Ph. D,, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Biliary drainage in KT
Record Dates: First submitted 2017-03-25; First posted 2017-04-07 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Cholangitis
Keywords: ERCP; PTBD; EBD; Cholangitis; Complication; Klatskin tumor
MeSH Terms: conditions — Cholangitis; Klatskin Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biliary drainage 1 (Experimental): Patients with advanced hilar cholangiocarcinoma need biliary drainage performed Endoscopic Retrograde Cholangiopancreatography (ERCP) drainage
  Interventions: Procedure: ERCP Drainage
- Biliary drainage 2 (Active Comparator): Patients with advanced hilar cholangiocarcinoma need biliary drainage performed percutaneous transhepatic biliary drainage(PTBD) drainage
  Interventions: Procedure: PTBD Drainage

INTERVENTIONS:
Procedure: ERCP Drainage — When advanced Klatskin Tumor patients need biliary drainage, they choose to perform endoscopic drainage after informed consent.
  Arms: Biliary drainage 1
Procedure: PTBD Drainage — When advanced Klatskin Tumor patients need biliary drainage, they choose to perform percutaneous transhepatic biliary drainage after informed consent.
  Arms: Biliary drainage 2

SUMMARY:
To investigate the biliary drainage-related cholangitis and other complications of percutaneous transhepatic biliary drainage (PTBD) in the management of Klatskin tumor (KT) compared with endoscopic biliary drainage (EBD).

DETAILED DESCRIPTION:
Operative treatment combined with preoperative biliary drainage (PBD) has been established as a safe management strategy for KT. Preoperative cholangitis was an independent risk factor for patients undergoing resection for KT. However, controversy exists regarding the preferred technique for PBD.

ELIGIBILITY:
Inclusion Criteria:

* Type II、III、IV Klatskin tumor patients;
* 18-90 years old

Exclusion Criteria:

* Unwillingness or inability to consent for the study;
* Coagulation dysfunction (INR> 1.3) and low peripheral blood platelet count(<50×109 / L) or using anti-coagulation drugs;
* Previous endoscopic sphincterectomy (EST) or endoscopic papillary balloon dilatation (EPBD);
* Any type of GI reconstruction;
* Combined with Mirizzi syndrome and intrahepatic bile duct stones;
* Preoperative coexistent diseases: acute pancreatitis, GI tract hemorrhage, severe liver disease, primary sclerosing cholangitis (PSC), septic shock;
* Biliary-duodenal fistula;
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Acute cholangitis | 2 weeks
  Acute cholangitis is defined if patients experienced abdominal pain, high fever, or chill after procedure in 2 weeks

SECONDARY OUTCOMES:
Abdominal pain | 2 weeks
  Pain score (scores:1-10)
Length of hospital stay | 6 months
  The total time of hospital stay
Overall procedure related complication rate | 6 months
  Pancreatitis, bleeding, perforation, seeding

CONTACTS AND LOCATIONS:
Overall Officials: Xun Li, M.D., Ph. D., Study Director — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ba Y, Yue P, Leung JW, Wang H, Lin Y, Bai B, Zhu X, Zhang L, Zhu K, Wang W, Meng W, Zhou W, Liu Y, Li X. Percutaneous transhepatic biliary drainage may be the preferred preoperative drainage method in hilar cholangiocarcinoma. Endosc Int Open. 2020 Feb;8(2):E203-E210. doi: 10.1055/a-0990-9114. Epub 2020 Jan 22. PMID 32010755